CLINICAL TRIAL: NCT02615171
Title: RELAX: A Mobile Application Suite Targeting Obesity and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Worcester Polytechnic Institute (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Sherry Pagoto, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H17-217; 1R01HL122302-01A1 (NIH)
Record Dates: First submitted 2015-11-19; First posted 2015-11-26 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Stress; Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive Dietary Self-Monitoring (Active Comparator): The intervention includes Facebook-delivered weight loss counseling and the use of MyFitnessPal, a comprehensive diet and exercise self-monitoring app. The intervention will last for 12 weeks. In addition to weight loss counseling in a private Facebook group, participants will be encouraged to use the self-monitoring app to enter everything they eat and do for exercise during the intervention period (12 weeks). Participants will receive a daily calorie goal directly from the app. Participants will receive a Fitbit scale to take their weight weekly and at assessments.
  Interventions: Behavioral: Comprehensive Dietary Self-Monitoring; Device: smartphone; Other: physical activity
- Simple Dietary Self-Monitoring (Active Comparator): The intervention includes Facebook-delivered weight loss counseling and the use of Slip Buddy, an app created by the investigative team that only requires users to record instances of overeating by hitting a single button and then indicate the overeating trigger and stress and hunger levels. The intervention will last for 12 weeks. In addition to the weight loss counseling, participants will be asked to use the Slip Buddy app during the intervention period (12 weeks). Participants will receive a Fitbit scale to take their weight weekly and at assessments.
  Interventions: Behavioral: Simple Dietary Self-Monitoring; Device: smartphone; Other: physical activity

INTERVENTIONS:
Behavioral: Comprehensive Dietary Self-Monitoring; Device: smartphone; Other: physical activity — The intervention includes Facebook-delivered weight loss counseling and the use of MyFitnessPal, a comprehensive diet and exercise self-monitoring app. The intervention will last for 12 weeks. In addition to weight loss counseling in a private Facebook group, participants will be encouraged to use the self-monitoring app to enter everything they eat and do for exercise during the intervention period (12 weeks). Participants will receive a daily calorie goal directly from the app. Participants will receive a Fitbit scale to take their weight weekly and at assessments.
  Arms: Comprehensive Dietary Self-Monitoring
Behavioral: Simple Dietary Self-Monitoring; Device: smartphone; Other: physical activity — Arm: Active Comparator: Simple Dietary Self-Monitoring he intervention includes Facebook-delivered weight loss counseling and the use of Slip Buddy, an app created by the investigative team that only requires users to record instances of overeating by hitting a single button and then indicate the overeating trigger and stress and hunger levels. The intervention will last for 12 weeks. In addition to the weight loss counseling, participants will be asked to use the Slip Buddy app during the intervention period (12 weeks). Participants will receive a Fitbit scale to take their weight weekly and at assessments.
  Arms: Simple Dietary Self-Monitoring

SUMMARY:
This research is being done is to evaluate the feasibility and acceptability of a novel weight loss mobile app that was designed to be less burdensome than traditional weight loss apps.

DETAILED DESCRIPTION:
Obesity and stress are highly comorbid and both increase risk for cardiovascular disease (CVD). Stress is associated with disinhibited eating, junk food consumption and low consumption of produce and whole grains. Both stress and stress-induced eating are not only associated with obesity but also predict worst outcomes in lifestyle interventions. Stress and stress-induced eating should be targeted in interventions to maximize weight loss; however, this makes for a very intensive intervention. Technology could be leveraged to reduce intervention burden.

In this trial investigators propose to compare the feasibility, usability, acceptability, and burden of an traditional weight loss app that includes diet and physical activity self-monitoring features to an app (Slip Buddy) we developed that focuses on self-monitoring of stress eating. With Slip Buddy, the user is just asked to track overeating episodes, indicating when they are triggered by stress. The majority of weight loss apps are burdensome to users by requiring them to self-monitor diet and exercise. They also ignore major barriers to weight loss, such as stress. This work moves the field forward by addressing user burden and an important barrier to weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Have a BMI of 27-45
* Currently use an Android smartphone
* Have cell phone connectivity at home and work
* Uses a smartphone every day

Exclusion Criteria:

* Under the age of 18 and over the age of 65;
* BMI under 27 or over 45;
* Not interested in losing weight;
* Does not currently own a smartphone;
* Smartphone type and/or version not meeting app requirements;
* No phone connectivity at home and work;
* Unable to walk unaided for ¼ mile without stopping;
* Has a condition that precludes dietary changes (i.e. ulcerative colitis, Crohn's disease, active diverticulitis, renal disease);
* On a medication affecting weight;
* Type 1 or 2 diabetes;
* Had gastric bypass surgery;
* Had or plans to have gastric bypass surgery during the study period;
* Pregnant/lactating;
* Has bipolar disorder, substance abuse, bulimia, or severe depression;
* Lost 5% or more body weight in the last 3 months;
* Has not experienced emotional eating over the last week;
* On medication affecting weight;
* Has concerns about being audiotaped;
* Prisoner;
* Unable to provide consent; or
* Non-English speaking

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

REFERENCES:
- [Derived] Pagoto S, Tulu B, Waring ME, Goetz J, Bibeau J, Divito J, Groshon L, Schroeder M. Slip Buddy App for Weight Management: Randomized Feasibility Trial of a Dietary Lapse Tracking App. JMIR Mhealth Uhealth. 2021 Apr 1;9(4):e24249. doi: 10.2196/24249. PMID 33792547

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After participants were initially screened, a telephone screening, webinar orientation and baseline survey was required prior to being randomized.
Period: Overall Study
Arm/Group | Comprehensive Dietary Self-Monitoring | Simple Dietary Self-Monitoring
Started | 32 | 32
Completed | 30 | 31
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Comprehensive Dietary Self-Monitoring | Simple Dietary Self-Monitoring | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.2 (12.3) | 39.5 (9.6) | 39.8 (11.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Selection of Gender: Male | 7 | 8 | 15
  Selection of Gender: Female | 24 | 24 | 48
  Selection of Gender: Transmasculine Nonbinary | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 28 | 31 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 28 | 27 | 55
  More than one race | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days App Used Over 12 Weeks
Description: App use was measured for each condition using either backend data from Slip Buddy or reviewing MyFitnessPal entries indicating use over each 24-hour period.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent of days app used
Arm/Group | Comprehensive Dietary Self-Monitoring | Simple Dietary Self-Monitoring
Number analyzed (Participants) | 32 | 32
percent of days app used | 57.5 (28.4) | 53.8 (31.3)

2. Primary Outcome: Usability
Description: Usability will be assessed using the System Usability Scale (SUS), a 10-item measure with 5-point Likert scale response options (Strongly Agree to Strongly Disagree). Scores are summed (0-40) then converted to a 0-100 scale, with higher scores indicating higher usability. Scores above 58 are considered above average, and scores above 80 are considered to indicate high usability where participants are likely to recommend the product to friends.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Dietary Self-Monitoring | Simple Dietary Self-Monitoring
Number analyzed (Participants) | 30 | 31
score on a scale | 76.3 (17.6) | 64.8 (16.5)
Statistical Analysis 1: Comparison: Comprehensive Dietary Self-Monitoring vs Simple Dietary Self-Monitoring; Test type: Other; p = 0.0106, t-test, 2 sided

3. Primary Outcome: Acceptability
Description: Acceptability was assessed with a single item at 12 weeks assessing perceived helpfulness of the assigned app: "Tracking my diet and exercise with MFP/slips with Slip Buddy was helpful" (responses on a 5-point Likert scale from strongly disagree to strongly agree). Acceptability was indicated by responses of agree or strongly agree.
Time Frame: 12 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Comprehensive Dietary Self-Monitoring | Simple Dietary Self-Monitoring
Number analyzed (Participants) | 30 | 31
percentage of participants | 77 | 39
Statistical Analysis 1: Comparison: Comprehensive Dietary Self-Monitoring vs Simple Dietary Self-Monitoring; Test type: Other; p = 0.0027, Chi-squared

4. Primary Outcome: Burden
Description: At 12 weeks, participants were asked how burdensome the task of using their assigned application was on a scale of 0-100, 0 being not at all burdensome and 100 being very burdensome.
Time Frame: 12 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Comprehensive Dietary Self-Monitoring | Simple Dietary Self-Monitoring
Number analyzed (Participants) | 30 | 31
units on a scale | 45.0 [10.0 to 60.0] | 30.0 [15.0 to 50.0]
Statistical Analysis 1: Comparison: Comprehensive Dietary Self-Monitoring vs Simple Dietary Self-Monitoring; Test type: Other; p = 0.7829, Wilcoxon rank sum test

5. Secondary Outcome: Percent Weight Change From Baseline to 12-Week Follow-Up
Description: A digital scale (Fitbit Aria) will be used to record weight. Percent weight change was calculated using weight at baseline and weight at 12-week follow-up. Missing values were calculated using last carry forward (LOCF).
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percent weight
Arm/Group | Comprehensive Dietary Self-Monitoring | Simple Dietary Self-Monitoring
Number analyzed (Participants) | 32 | 32
percent weight | -3.6 (4.9) | -3.0 (4.5)

6. Secondary Outcome: Change in Perceived Stress From Baseline to 12-Week Follow-Up
Description: The Perceived Stress Scale is a 14-item measure of perceived stress. Scores range from 0-56, higher scores indicate higher perceived stress.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Comprehensive Dietary Self-Monitoring | Simple Dietary Self-Monitoring
Number analyzed (Participants) | 30 | 31
score on a scale | 2.8 (9.1) | 2.5 (6.8)

7. Secondary Outcome: Change in Emotional Eating From Baseline to 12-Week Follow-Up
Description: Three-Factory Eating Inventory is an 18-item measure and the emotional eating subscale consists of 3 items on a 4-point Likert scale. The score is derived by a multi-step equation. The range of scores for this subscale is 0-100, higher scores indicate higher emotional eating.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: change in score from baseline 12 weeks
Arm/Group | Comprehensive Dietary Self-Monitoring | Simple Dietary Self-Monitoring
Number analyzed (Participants) | 30 | 31
change in score from baseline 12 weeks | -1.1 (25.5) | -9.9 (25.1)

ADVERSE EVENTS:
Time Frame: Adverse events were collected over the period of 12 weeks.
Description: Adverse events were assessed during follow-up as well as documented when participants reported them during the intervention. Pregnancy was only assessed with female participants.
Arm/Group | Comprehensive Dietary Self-Monitoring | Simple Dietary Self-Monitoring
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 5/32 | 5/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Comprehensive Dietary Self-Monitoring (N=32) | Simple Dietary Self-Monitoring (N=32)
Weight Gain (General disorders) | 1 (1) | 1 (1)
Injury unrelated to exercise (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1/24 (1) | 1/24 (1) — Assessed in females only
Flu (Immune system disorders) | 1 (1) | 0 (0)
Pulled Muscle During Exercise (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT02615171/Prot_001.pdf
  • Statistical Analysis Plan (2020-10-29): https://cdn.clinicaltrials.gov/large-docs/71/NCT02615171/SAP_002.pdf
  • Informed Consent Form (2019-08-31): https://cdn.clinicaltrials.gov/large-docs/71/NCT02615171/ICF_003.pdf